CLINICAL TRIAL: NCT00096954
Title: A Prospective, Randomized, Double-Blind Study of the Efficacy of Omalizumab (Xolair) in Atopic Asthmatics With Good Lung Capacity Who Remain Difficult to Treat (EXACT)
Acronym: EXACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q2982g
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Omalizumab (Xolair); Atopic Asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Omalizumab (Experimental): Omalizumab (Xolair) administered in this study was either a minimum of 0.008 mg/kg/IgE [IU/mL] every 2 weeks or a minimum of 0.016 mg/kg/IgE [IU/mL] every 4 weeks.
  Interventions: Drug: omalizumab (Xolair)
- Placebo (Placebo Comparator): Placebo administered in this study was either a minimum of 0.008 mg/kg/IgE [IU/mL] every 2 weeks or a minimum of 0.016 mg/kg/IgE [IU/mL] every 4 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: omalizumab (Xolair) — Omalizumab (Xolair) was administered subcutaneously every 2 or 4 weeks. The dose (mg) and dosing frequency were determined by serum total IgE level (IU/mL), measured before the start of treatment, and body weight (kg). Assignment of the study drug dose was determined by using the study drug-dosing table. Doses of > 150 mg were divided among more than one injection site to limit injections to no more than 150 mg per site.
  Arms: Omalizumab
Drug: placebo — The dose of placebo consisting of sucrose, L-histidine, L-histidine hydrochloride monohydrate, and polysorbate 20 was administered by subcutaneous injection every 2 or 4 weeks.
  Arms: Placebo

SUMMARY:
This was a multicenter, parallel-group, double-blind, randomized, placebo-controlled study that enrolled 333 subjects. These subjects were 12-75 years old with atopic asthma, had elevated serum total Immunoglobulin E (IgE), had a baseline forced expiratory volume in 1 second (FEV1) ≥ 80% predicted, and were on inhaled corticosteroids with or without other controller asthma medications (e.g., long-acting β2-agonists [LABAs], leukotriene receptor antagonist [LTRA], or immunotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Have a documented history of asthma as well as evidence of ≥ 12% reversibility of FEV1. Evidence of ≥ 12% reversibility of FEV1 may be obtained by any one of the following measures: 1) Documentation of ≥ 12% reversibility of FEV1 after albuterol administration at any time during the preceding 24 months; 2) Documentation of ≥ 12% improvement in FEV1 with two separate measurements obtained within a 4-week period surrounding an asthma exacerbation during the preceding 24 months; 3) Demonstration of ≥ 12%reversibility of FEV1 after albuterol administration at the time of screening
* Have baseline FEV1 ≥ 80% predicted normal value prior to randomization
* Have a positive skin test (diameter of wheal ≥ 3 mm vs. control) or in vitro radioallergosorbent test (RAST(R)) or ImmunoCap(R) to one relevant perennial aeroallergen such as cat or house dust mites documented within the previous year
* Be receiving at least an inhaled corticosteroid dosage of fluticasone dry powder inhaler (DPI) ≥ 200 ug/day or equivalent ex-valve dose during the 12 weeks prior to the screening visit
* During the 4-week run-in period prior to randomization, demonstrate evidence of inadequate asthma symptom control despite inhaled corticosteroids with or without other controller asthma medications (e.g., LABA, LTRA, immunotherapy). Inadequate asthma symptom control is defined as at least one of the following reported on the subject diary card during the 4-week run-in period: Daytime asthma symptoms as a score of ≥ 1 (scale of 0-4) on at least 20 of 28 days (missing data to be treated as a day with no symptoms) and a mean symptom score of ≥ 1.5 (mean will be calculated based on only data supplied; missing values will not be considered) or Nighttime awakening because of asthma symptoms (more than 4 times during the 4-week run-in period)
* Meet the study drug-dosing table eligibility criteria (serum baseline IgE level ≥ 30 to ≤ 1300 IU/mL and body weight ≥ 20 to ≤ 150 kg)
* If a female of childbearing potential, use an effective method of contraception (in the opinion of the investigator) to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of their participation in the study

Exclusion Criteria:

* Have received chronic systemic corticosteroids (oral or intravenous) within 3 months or have received a burst of oral corticosteroids within the last 2 weeks prior to screening
* Have received Xolair therapy at any time within 12 months prior to screening
* Are pregnant or lactating
* Have a known hypersensitivity to any ingredients of Xolair, including excipients (sucrose, histidine, polysorbate 20)
* Have a lifetime history of smoking > 10-pack years
* Have active lung disease other than asthma (e.g., chronic bronchitis, emphysema, cystic fibrosis, chronic obstructive pulmonary disease)
* Have a history of upper respiratory infection or lower respiratory infection within the 30 days prior to randomization
* Have a diagnosis of aspirin or nonsteroidal anti-inflammatory drug-induced asthma
* Have taken immunosuppressants or other investigational drugs within the 30 days prior to screening
* Have a significant medical illness other than asthma

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Rosen, MD, PhD, Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab (Xolair) | Placebo
Started | 159 | 174
Received Study Drug | 157 | 171
Completed | 135 | 154
Not Completed | 24 | 20
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Physician Decision | 1 | 1
Not completed — Sponsors Decision | 1 | 1
Not completed — Pregnancy | 1 | 1
Not completed — Initiation of immunotherapy | 1 | 0
Not completed — Non-compliance | 0 | 3
Not completed — Lost to Follow-up | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Placebo: The dose of placebo was administered by subcutaneous injection every 2 or 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Omalizumab (Xolair) | Placebo | Total
Number analyzed (Participants) | 157 | 171 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (14.7) | 38.1 (15.1) | 37.1 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristic numbers reflect the number of participants who received at least one dose of drug. Two participants in the Xolair group and three participants in the placebo group were not dosed.
  Participants
    Female | 110 | 116 | 226
    Male | 47 | 55 | 102

OUTCOME MEASURES:

1. Primary Outcome: Rate of Asthma Exacerbations Over the 24 Week Treatment Period
Description: A protocol-defined asthma exacerbation was a worsening of asthma requiring treatment with oral or intravenous corticosteroid burst and/or a doubling of the baseline inhaled corticosteroids (ICS) dose for at least 3 days.
  The rate of protocol-defined asthma exacerbations, normalized by subject-time at risk and computed over the 24 week treatment period in each treatment group.
Time Frame: Start of treatment to 24 weeks
Population: Modified Intent-to-Treat - All randomly assigned patients who received at least 1 dose of study drug (omalizumab or placebo).
Measure: Number; unit: exacerbations per 24 patient-week period
Arm/Group | Omalizumab (Xolair) | Placebo
Number analyzed (Participants) | 157 | 171
exacerbations per 24 patient-week period | 0.205 | 0.258

2. Secondary Outcome: Number of Participants Experiencing One or More Protocol-defined Asthma Exacerbations During the Treatment Period
Description: The number of patients reporting one or more protocol-defined asthma exacerbations during the 24 week treatment period. A protocol-defined asthma exacerbation was a worsening of asthma requiring treatment with oral or intravenous corticosteroid burst and/or a doubling of the baseline inhaled corticosteroids (ICS) dose for at least 3 days.
Time Frame: Start of treatment to 24 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Omalizumab (Xolair) | Placebo
Number analyzed (Participants) | 157 | 171
participants | 24 | 33

3. Secondary Outcome: Change From Baseline in Nocturnal and Daytime Asthma Symptom Scores at Week 24
Description: The daytime asthma symptom score assessed the symptoms: shortness of breath, chest discomfort, wheezing, and cough over the previous 24 hour period on a scale of 0(no symptoms) to 4(marked discomfort).
  The nocturnal asthma score was the patient's response to:How did you sleep last night? rated on a scale of 0(no problems) to 4(difficulty sleeping;rescue medicine used).
  Scores were collected daily. Change from Baseline (mean of last 28 days prior to first dosing date) at Week 24 (mean of last 28 days prior to week 24 visit).
  A negative change from baseline score indicates improvement.
Time Frame: Baseline and 24 weeks
Population: Modified Intent-to-Treat. Patients with missing Asthma Symptom Score data at week 24 were excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omalizumab (Xolair) | Placebo
Number analyzed (Participants) | 132 | 154
score on a scale
  Daytime | -0.73 (0.72) | -0.67 (0.72)
  Nocturnal | -0.48 (0.77) | -0.49 (0.67)

4. Secondary Outcome: Relative Percent Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 24
Description: Spirometry was used to assess FEV1. All spirometry measurements were performed in accordance with the American Thoracic Society (ATS) guidelines.
  The relative percent change from baseline in forced expiratory volume (liters) in one second (FEV1) was calculated at week 24 using the formula: (FEV1 at week 24 - FEV1 at baseline) / FEV1 at baseline * 100 for each treatment group.
Time Frame: Baseline and 24 weeks
Population: Modified Intent-to-Treat. Patients with missing FEV1 data at either baseline or week 24 were excluded.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Omalizumab (Xolair) | Placebo
Number analyzed (Participants) | 135 | 153
percent change | 4.15 (21.53) [1.23 to 8.39] | -0.75 (11.90) [1.23 to 8.39]

ADVERSE EVENTS:
Time Frame: From first dosing date to 30 days after last dosing date, or the last day on study, whichever is earlier. (Up to 29.3 weeks)
Arm/Group | Omalizumab (Xolair) | Placebo
Serious Adverse Events (participants affected / at risk) | 4/157 | 6/171
Other Adverse Events (participants affected / at risk) | 36/157 | 56/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (Xolair) (N=157) | Placebo (N=171)
Esophageal perforation (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abortion induced (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (Xolair) (N=157) | Placebo (N=171)
upper respiratory tract infection (Infections and infestations) | 15 | 17
sinusitis (Infections and infestations) | 11 | 16
nasopharyngitis (Infections and infestations) | 9 | 16
headache (Nervous system disorders) | 7 | 10

LIMITATIONS AND CAVEATS:
This is a stand-alone study to fulfill one of the post-marketing commitments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.